CLINICAL TRIAL: NCT04667650
Title: Use of Nomogram for Predictions of Ocular Mysathenia Gravis Generalization
Brief Title: Ocular Mysathenia Gravis Generalization
Acronym: MYASTEN
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Principal Investigator, Amélie Yavchitz, Dr Amélie Yavchitz, Fondation Ophtalmologique Adolphe de Rothschild
Other Study IDs: CE_20161027_22_AGN
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Ocular Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Use of nomogram for predictions of Ocular Mysathenia Gravis generalization — The outcome measure was time to Myasthenia gravis generalization. The explanatory variables were age at onset, sex, first-year anti-acetylcholinereceptor antibody positivity, repetiting nerve stimulation showing electromyogram decrement and steroid use. Kaplan-Meier survival estimations, descriptive and multivariate Cox model analyses were computed. A nomogram combining explanatory vraiables was used to establish a score to predict the probability of OMG generalization.

SUMMARY:
Secondary ocular myasthenia gravis (OMG) generalization represents a pejorative evolution and no validated generalization prevention strategy exists. The aim of this observational study was to determine the percentage of patients with OMG generalization and identify factors predictive of that pejorative evolution. Data from patients with OMG registered in the Fondation Hospital A. de Rothschild database between January 1990 and January 2017 were collected. Among the 183 patients registered in this database, 151 patients with available informations were analyzed.

ELIGIBILITY:
Inclusion Criteria:

- Patients with OMG diagnosis and its generalization who consulted between January 1990 to January 2017 at Fondation Hospital Adolphe de Rothschild and registered in the database

Exclusion Criteria:

- OMG differential diagnoses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with OMG diagnosis and its generalization who consulted between January 1990 to January 2017 at Fondation Hospital Adolphe de Rothschild and registered in the database
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Time to myasthenia gravis generalization | 1 year
  Kaplan-meier survival estimations, descriptive and multivariate Cox model analyses were computed (age at onset, first year anti-acetylcholine receptor antibody positivity, electromyogram decrement, steroid use).

CONTACTS AND LOCATIONS:
Locations (1):
- Antoine GUEGUEN, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided